CLINICAL TRIAL: NCT00413049
Title: A Multi-national, Multicenter, Double-blind, Double-dummy, Randomized, Active-controlled, Parallel Study Comparing the Efficacy and Safety of Valsartan/Amlodipine 80/5 mg to Amlodipine 5 mg Alone Once Daily in Patients With Mild to Moderate Essential Hypertension Not Adequately Controlled With Amlodipine 5 mg Monotherapy
Brief Title: Efficacy/Safety of Valsartan Plus Amlodipine and Amlodipine Alone in Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis Medical Director, Novartis Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAA489A2315
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Results first posted 2011-02-08 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
Keywords: Hypertension, valsartan, amlodipine, high blood pressure
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Valsartan/amlodipine 80/5 mg (Experimental)
  Interventions: Drug: Valsartan/amlodipine 80/5 mg
- Amlodipine 5 mg (Active Comparator)
  Interventions: Drug: Amlodipine 5 mg

INTERVENTIONS:
Drug: Valsartan/amlodipine 80/5 mg — 1 valsartan/amlodipine 80/5 mg tablet and 1 placebo capsule matching amlodipine 5 mg to be taken with water at approximately 8:00 a.m. once daily, except on the morning of every scheduled study visit, when study drug was taken after the completion of all other study procedures.
  Arms: Valsartan/amlodipine 80/5 mg
Drug: Amlodipine 5 mg — 1 amlodipine 5 mg capsule and 1 placebo tablet matching valsartan/amlodipine 80/5 mg to be taken with water at approximately 8:00 a.m. once daily, except on the morning of every scheduled study visit, when study drug was taken after the completion of all other study procedures.
  Arms: Amlodipine 5 mg

SUMMARY:
This study will evaluate the safety and efficacy of the fixed combination of valsartan/amlodipine in adult patients with mild to moderate hypertension

ELIGIBILITY:
Inclusion criteria

* Male or female outpatients ≥ 18 years and < 86 years
* Patients with essential hypertension measured by calibrated mercury sphygmomanometer (preferred) or an aneroid device if a mercury sphygmomanometer was not available.
* At Visit 1, patients not treated with antihypertensive medications had to have a MSDBP of ≥ 95 mmHg and < 110 mmHg; those patients treated with antihypertensive medication had to have a MSDBP of < 110 mmHg.
* At Visit 2, patients must have a MSDBP of ≥ 95 mmHg but < 110 mmHg.
* At Visit 3, patients must have a MSDBP of ≥ 90 mmHg and < 110 mmHg.
* Patients who were eligible and able to participate in the study, and who consented to do so after the purpose and nature of the investigation had been clearly explained to them (written informed consent).

Exclusion criteria

* Severe hypertension (MSDBP ≥ 110 mmHg and/or MSSBP ≥ 180 mmHg).
* In cases where the patient was on more than one antihypertensive drug whether in fixed or free combination, the investigator considered the efficacy and strength of each active ingredient in order to determine if the patient could be safely removed from their antihypertensive treatment.
* Known or suspected contraindications, including history of allergy or hypersensitivity to angiotensin receptor blockers (ARB), calcium channel blockers (CCB), or to drugs with similar chemical structures.
* Administration of any agent indicated for the treatment of hypertension after Visit 1 with the exception of those agents that required tapering down.
* Inability to discontinue all prior antihypertensive medications safely for a maximum period of up to 28 days prior to Visit 2, as required by the protocol.
* History of hypertensive encephalopathy, cerebrovascular accident or transient ischemic attack, myocardial infarction or all types of revascularization.
* Malignant hypertension.
* All patients with Type 1 diabetes mellitus and those patients with Type 2 diabetes mellitus who were not well controlled based on the investigator's clinical judgment. Patients being treated for diabetes mellitus had to have satisfactory metabolic control. Type 2 diabetic patients taking oral anti-diabetic medication had to be on a stable dose for at least 4 weeks prior to Visit 1.
* Pregnant or nursing (lactating) women, where pregnancy was defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 5 mIU/ml).
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precluded intercourse with a male partner and women whose partners had been sterilized by vasectomy or other means, UNLESS they met the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) levels > 40 mIU/m or 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy OR were using one or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation, vasectomy), and double-barrier methods (any double combination of: intra-uterine device [IUD], male or female condom with spermicidal gel, diaphragm, sponge, cervical cap). Acceptable methods of contraception included total abstinence at the discretion of the investigator in cases where the age, career, lifestyle, or sexual orientation of the patient ensured compliance. Reliable contraception had to be maintained throughout the study and for 7 days after study drug discontinuation. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal were not acceptable methods of contraception. Hormonal contraceptive use was disallowed.
* History of heart failure Grade II-IV according to the New York Heart Association (NYHA) classification.
* Second or third degree heart block with or without a pacemaker.
* Concomitant potentially life threatening arrhythmia or symptomatic arrhythmia.
* Angina pectoris of any type, including unstable angina pectoris.
* Clinically significant valvular heart disease.
* Evidence of a secondary form of hypertension, including but not limited to any of the following: coarctation of the aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing disease, pheochromocytoma, polycystic kidney disease.
* Known moderate or malignant retinopathy, defined as: moderate (retinal signs of hemorrhage, microaneurysm, cotton-wool spot, hard exudates, or a combination thereof) or malignancy (signs of moderate retinopathy plus swelling of the optic disk).
* Evidence of hepatic disease as determined by any one of the following: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values greater than two times the upper limit of normal at Visit 1, a history of hepatic encephalopathy, a history of esophageal varices, or a history of a portocaval shunt.
* Evidence of renal impairment as determined by anyone of the following: serum creatinine > 1.5 times the upper limit of normal at Visit 1, a history of dialysis, or a history of nephrotic syndrome.
* History of clinically significant allergies including asthma, and/or multiple drug allergies.
* Any surgical or medical condition with the potential to significantly alter the absorption, distribution, metabolism, or excretion of any drug including but not limited to any of the following: history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, gastric bypass, gastric stapling, or gastric banding, currently active or active inflammatory bowel syndrome within 12 months prior to Visit 1, currently active gastritis, ulcers, or gastrointestinal/rectal bleeding, or urinary tract obstruction regarded as clinically meaningful by the investigator.
* Any surgical or medical condition, which in the opinion of the investigator or the Novartis monitor, placed the patient at higher risk from his/her participation in the study, or were likely to prevent the patient from complying with the requirement of the study or completing the trial period.
* Volume depletion based on the investigator's clinical judgment using vital signs, skin turgor, moistness of mucous membranes, and laboratory values.
* Any chronic inflammatory condition requiring chronic anti-inflammatory therapy.
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there was evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
* History of drug of alcohol abuse within the last 2 years.
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever was longer.
* Inability to communicate and comply with all study requirements including the unwillingness or inability to provide informed consent.
* Persons directly involved in the execution of this protocol.
* History of non-compliance to medical regimens, or unwillingness to comply with the study protocol.
* Currently taking prohibited concomitant medications(s) listed and inability/unwillingness to discontinue them for the entire study period.
* Any severe, life-threatening disease within the past five years.
* Arm circumference > 42 cm for patients participating in ambulatory blood pressure monitoring (ABPM).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Sponsor GmbH
Locations (12):
- China (12):
  - China-Japan Friendship Hospital, Beijing
  - People's hospital affiliated Beijing University, Beijing
  - The third Xiangya hospital of central south University, Changsha
  - The first hospital affiliated the third military Medical University, Chongqing
  - The third hospital affiliated the third military Medical University, Chongqing
  - Union hospital affiliated Fujian medical University, Fuzhou
  - The first hospital affiliated Fujian medical University, Fuzhou
  - The second hospital affiliated Jiangxi medical school, Nanchang
  - Institute of Hypertension, Ruijin Hospital, Shanghai
  - Zhongshan hospital affiliated Fudan University, Shanghai
  - The sixth people's hospital of Shanghai, Shanghai
  - The first hospital affiliated school of medical of Xi'an Jiaotong University, Xi'an

REFERENCES:
- [Derived] Ke Y, Zhu D, Hong H, Zhu J, Wang R, Cardenas P, Zhang Y. Efficacy and safety of a single-pill combination of amlodipine/valsartan in Asian hypertensive patients inadequately controlled with amlodipine monotherapy. Curr Med Res Opin. 2010 Jul;26(7):1705-13. doi: 10.1185/03007995.2010.487391. PMID 20469975

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients in the valsartan/amlodipine group were excluded from the intent-to-treat population used for the efficacy analyses for having no post-baseline efficacy assessment.
Period: Overall Study
Arm/Group | Valsartan/Amlodipine 80/5 mg | Amlodipine 5 mg
Started | 349 | 349
Completed | 325 | 331
Not Completed | 24 | 18
Not completed — Adverse Event | 10 | 8
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Lost to Follow-up | 2 | 3
Not completed — Protocol Violation | 3 | 1
Not completed — Subject no longer requires study drug | 0 | 1
Not completed — Abnormal laboratory value(s) | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan/Amlodipine 80/5 mg | Amlodipine 5 mg | Total
Number analyzed (Participants) | 347 | 349 | 696
Age Continuous [Mean (Standard Deviation); unit: years] | 53.4 (9.7) | 54.2 (9.1) | 53.8 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 109 | 243
  Male | 213 | 240 | 453

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Baseline to End of Study (Week 8)
Description: Blood pressure (BP) was measured with a calibrated aneroid or mercury sphygmomanometer. The arm in which the highest sitting diastolic BP was found at study entry was used for all subsequent readings. At each visit, after the patient was in a sitting position for five minutes, systolic/diastolic BP was measured 3 times at 1-2-minute intervals. The mean of the 3 measurements was calculated. A negative change score indicates lowered BP.
Time Frame: Baseline to end of study (Week 8)
Population: Intent-to-Treat (ITT): All randomized patients who had baseline and at least one post-baseline efficacy measurement, ie, any post-baseline measurement of primary or secondary efficacy variables. For patients who did not complete the Week 8 assessment, a last observation carried forward (LOCF) approach was used.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 80/5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 347 | 349
mmHg | -9.7 (0.42) | -7.1 (0.42)

2. Secondary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) From Baseline to End of Study (Week 8)
Description: as for outcome 1
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Valsartan/Amlodipine 80/5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 347 | 349
mmHg | -11.4 (0.61) | -7.4 (0.60)

3. Secondary Outcome: Percentage of Patients Achieving a Diastolic Response at the End of the Study (Week 8)
Description: A patient achieved a diastolic response if their msDBP < 90 mmHg at Week 8 or they had a ≥ 10 mmHg decrease in msDBP compared to baseline at the end of the study (Week 8). Blood pressure (BP) was measured with a calibrated aneroid or mercury sphygmomanometer. The arm in which the highest sitting diastolic BP was found at study entry was used for all subsequent readings. At each visit, after the patient was in a sitting position for five minutes, systolic/diastolic BP was measured 3 times at 1-2-minute intervals. The mean of the 3 measurements was calculated.
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan/Amlodipine 80/5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 347 | 349
Percentage of patients | 79.3 | 66.8

4. Secondary Outcome: Percentage of Patients Achieving Diastolic Control at the End of the Study (Week 8)
Description: A patient achieved diastolic control if their msDBP < 90 mmHg at the end of the study (Week 8). Blood pressure (BP) was measured with a calibrated aneroid or mercury sphygmomanometer. The arm in which the highest sitting diastolic BP was found at study entry was used for all subsequent readings. At each visit, after the patient was in a sitting position for five minutes, systolic/diastolic BP was measured 3 times at 1-2-minute intervals. The mean of the 3 measurements was calculated.
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan/Amlodipine 80/5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 347 | 349
Percentage of patients | 75.5 | 64.5

5. Secondary Outcome: Percentage of Patients Achieving Overall Control at the End of the Study (Week 8)
Description: A patient achieved overall control if the msSBP/msDBP < 140/90 mmHg at the end of the study (Week 8). Blood pressure (BP) was measured with a calibrated aneroid or mercury sphygmomanometer. The arm in which the highest sitting diastolic BP was found at study entry was used for all subsequent readings. At each visit, after the patient was in a sitting position for five minutes, systolic/diastolic BP was measured 3 times at 1-2-minute intervals. The mean of the 3 measurements was calculated.
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Valsartan/Amlodipine 80/5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 347 | 349
Percentage of patients | 69.2 | 57.6

6. Secondary Outcome: Change in 24-hour Mean Ambulatory Diastolic and Systolic BP From Baseline at the End of the Study (Week 8)
Description: Two 24 hour ambulatory blood pressure monitoring (ABPM) evaluations were performed, one at baseline prior to randomization and one at Week 8 (end of study), in a subset of the intent-to-treat population of patients. For each evaluation, the ABPM device was attached to the non-dominant arm of the patient. A correlation was made between the ABPM device readings and measurements taken with a mercury sphygmomanometer and stethoscope. Following the correlation procedure, BP was measured at study specified intervals. A negative change score indicates lowered BP.
Time Frame: Baseline to end of study (Week 8)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Valsartan/Amlodipine 80/5 mg | Amlodipine 5 mg
Number analyzed (Participants) | 41 | 41
mmHg
  Diastolic BP | -6.3 (5.85) | 0.3 (5.82)
  Systolic BP | -7.3 (7.62) | -0.2 (8.64)

ADVERSE EVENTS:
Arm/Group | Valsartan/Amlodipine 80/5 mg | Amlodipine 5 mg
Serious Adverse Events (participants affected / at risk) | 4/349 | 2/349
Other Adverse Events (participants affected / at risk) | 0/349 | 0/349
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan/Amlodipine 80/5 mg (N=349) | Amlodipine 5 mg (N=349)
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.